CLINICAL TRIAL: NCT06958965
Title: Effects of Resistance Exercise Training on Vascular Function and Physical Performance in Postmenopausal Women
Brief Title: Resistance Exercise Training on Vascular and Physical Function in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NYCU114053AE
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Postmenopausal Women
Keywords: exercise; cardiovascular diseases; arteries; arterial compliance; hormones; estrogen
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects of Resistance Exercise Training on Vascular Function and Physical Performance in Postmenopau (Experimental): This study involved a 12-week group-based resistance training program, with two sessions per week, each lasting 90 to 120 minutes. The exercise intensity targeted 40-70% of participants' one-repetition maximum (1RM) or a moderate level (approximately a score of 3 on the Modified Borg RPE scale). Equipment used included dumbbells, kettlebells, grip rings, body bars, resistance bands, step platforms, and sandbags, following a three-phase structured exercise model.
  Interventions: Other: Resistance exercise training
- Control (No Intervention): Participants in the control group did not undergo any resistance training intervention and were advised to continue their usual daily routines, dietary patterns, and prescribed medications throughout the study period.

INTERVENTIONS:
Other: Resistance exercise training — The total duration of the training was 12 weeks, with a frequency of two sessions per week. Each session lasted approximately 90 to 120 minutes. The exercise intensity was set at 40-70% of the participants' one-repetition maximum (1RM), or adjusted based on the Modified Borg Rating of Perceived Exertion (RPE), targeting a moderate intensity level (approximately a score of 3).
  Other Names: resistance training
  Arms: Effects of Resistance Exercise Training on Vascular Function and Physical Performance in Postmenopau

SUMMARY:
Postmenopausal women often face risks of vascular dysfunction and muscle deterioration due to estrogen deficiency. These changes significantly increase the risk of cardiovascular disease and mortality. Previous studies have shown a significant positive correlation between vascular endothelial function and muscle strength. Moreover, muscle strength is a stronger predictor of mortality than muscle mass and is closely associated with the maintenance of functional independence in daily life. However, studies investigating the effects of whole-body progressive resistance training on vascular function and physical performance in postmenopausal women remain limited. This study aims to examine changes in vascular function and muscle strength in postmenopausal women following a whole-body progressive resistance training program.

ELIGIBILITY:
Inclusion Criteria:

Participants were eligible for the study if they met the following criteria:

1. Postmenopausal women aged between 55 and 70 years;
2. Body mass index (BMI) less than 30 kg/m²;
3. At least one year since menopause;
4. Able to live independently in the community;
5. Able to communicate independently in Mandarin or Taiwanese.

Exclusion Criteria:

Participants were excluded if they met any of the following conditions:

1. Acute musculoskeletal injuries within the past month (e.g., acute inflammation, fractures, sprains, contusions, or joint implants);
2. Diagnosed central or peripheral nervous system disorders affecting exercise participation (e.g., stroke, dementia, Parkinson's disease, autonomic dysfunction);
3. History of serious cardiac conditions within the past six months (e.g., coronary stenting, pacemaker implantation, peripheral or cerebral vascular reconstruction);
4. Presence of peripheral vascular diseases (e.g., peripheral artery disease, venous thrombosis);
5. Hormone therapy within the past six months;
6. Currently taking beta-blockers, anti-inflammatory drugs, or anticoagulant medications;
7. Currently participating in any other structured exercise training programs.

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated dilation-endothelial function | Change from baseline at 12 weeks
  During the test, participants were instructed to remain in a supine position with the shoulder abducted to 90 degrees and the palm facing upward. A friction-reducing sleeve and a sphygmomanometer cuff were placed on the distal part of the non-dominant forearm. The cuff inflation pressure was set at least 50 mmHg above the systolic blood pressure measured from the dominant arm and maintained for 5 minutes. Immediately after the 5-minute occlusion period, the cuff was rapidly deflated, and the brachial artery diameter was continuously monitored for up to 3 minutes to capture post-deflation vascular changes.
Brachial-ankle plus wave velocity (baPWV)-arterial stiffness | Chang from baseline at 12 weeks
  A non-invasive assessment of arterial stiffness was conducted using an arterial stiffness device based on pulse wave velocity (PWV) measurement. During the test, participants were instructed to lie in a relaxed supine position in a quiet environment. Four blood pressure cuffs were placed on both arms and both ankles. The measurements from the left and right sides were averaged for analysis.The PWV was calculated using the following formula:
  PWV = Distance / Pulse Transit Time

SECONDARY OUTCOMES:
Hand grip strength- muscle strength | Change from baseline at 12 weeks
  Participants were instructed to stand with their feet shoulder-width apart, with elbows fully extended and slightly abducted at approximately 45 degrees. They were asked to apply maximum grip strength and hold for 3 to 4 seconds. Each hand was tested three times, with a 10- to 15-second rest between trials. Both hands were tested, and the highest value from each hand was recorded for analysis.
Five-repetition maximum test (5RM) | Change from baseline at 12 weeks
  In this study, exercise intensity was estimated using the five-repetition maximum (5RM) test to predict the one-repetition maximum (1RM). Given that the target population consisted of middle-aged and older postmenopausal women, the 5RM test was selected to reduce the risk of injury and enhance participant motivation.
  The predicted 1RM was calculated using the formula proposed by LeSuer et al.:
  1RM = body weight × (1 + 0.0333 × number of repetitions)
Body Composition | Change from baseline at 12 weeks
  Skeletal muscle mass index (SMI) of the limbs was assessed using multifrequency bioelectrical impedance analysis (MF-BIA; InBody 270, Tokyo, Japan). During the test, participants stood barefoot on the marked footplate positions with their arms relaxed and slightly abducted, placing their thumbs on the designated sensors. Each measurement lasted approximately 10 to 15 seconds while maintaining a standing posture.
Perceived Exertion | Change from baseline at 12 weeks
  This study utilized the Chinese version of the Modified Borg Rating of Perceived Exertion (RPE) scale to assess participants' subjective perception of effort. The scale ranges from 0 to 10, where a score of 0 indicates no exertion at all.
International Physical Activity Questionnaire (IPAQ) - Taiwan Physical Activity Questionnaire (Short Form) | Change from baseline at 12 weeks
  The IPAQ is a self-reported instrument assesses the time spent in the past 7 days on activities including work, housework, gardening/balcony work, commuting, leisure, and exercise. Total time spent per week is multiplied by the metabolic equivalent (MET) and summed to present the total MET-minutes per week. Physical activity intensity is classified into walking (3.3 METs), moderate (4.0 METs), and vigorous (8.0 METs).
Short Physical Performance Battery (SPPB) | Change from baseline at 12 weeks
  This assessment consisted of three components to evaluate lower extremity function. First, the standing balance test required participants to maintain balance in three stances-feet together, semi-tandem, and full tandem-for up to 10 seconds each. Second, the gait speed test measured the time it took participants to walk 4 meters at their usual pace, reflecting their walking speed. Third, the chair stand test assessed lower limb muscle strength by recording the time needed to complete five consecutive sit-to-stand movements with arms crossed over the chest. These tests collectively provided an objective measure of physical performance.
3-Meter Walk Test | Change from baseline at 12 weeks
  This test is used to assess lower limb strength, balance, gait, and functional mobility in older adults. At the start of the test, the participant sits on a chair with a backrest, placing both hands on their thighs. Upon instruction, the participant stands up, walks to a marker placed 3 meters away, turns around the marker, walks back, and sits down again. The test is performed at the fastest safe speed.
30-Second Chair Stand Test: | Change from baseline at 12 weeks
  While seated on a chair of standard height with feet flat on the floor, participants are instructed to cross their arms over their chest. Upon the start of the test, they repeatedly stand up and sit down as many times as possible within 30 seconds. The total number of completed repetitions is recorded.